CLINICAL TRIAL: NCT00763282
Title: Self-Management to Prevent Ulcers in Veterans With Spinal Cord Injury
Brief Title: Self-Management to Prevent Ulcers in Veterans With SCI (Spinal Cord Injury)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIR 06-203
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-10

CONDITIONS: Pressure Ulcers; Spinal Cord Injuries
Keywords: Spinal cord injuries; Pressure ulcers; Health behavior; self management; Rehabilitation; Outcome assessment; QUERI; Veterans
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries; Health Behavior | interventions — Self-Management; Motivational Interviewing; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SM+MI (Experimental): Self Management (SM) + Motivational Interviewing (MI). Self Management and Motivational Interviewing (SM+MI) participants were assigned to both a self-management and motivational interview group. Motivational Interviewing (MI) is an evidence-based form of counseling to help individuals to engage in behavior change. Self Management (SM) consists of: 1) on-site decisional support to promote provider adherence to ulcer management guidelines, 2) enhanced, interactive PrU education, 3) chronic disease self-management skill building via telephone based groups, 4) proactive care management using MI to support ongoing self-management activities, and 5) distance technology.
  Interventions: Behavioral: Self Management (SM); Behavioral: Motivational Interviewing (MI)
- ED (Active Comparator): Education (ED). An education control intervention (ED) designed to be a credible intervention that is comparable to the SM will control for potential effects of natural history/time, treatment dosing, measurement processes, attention, the non-specific effects of therapeutic alliance, social support, and of receiving a manualized treatment with specific therapist procedures. The ED intervention will differ only in that subjects will not be instructed in any specific problem solving, self-monitoring, or SM techniques, with the exception of encouraging them to become informed consumers of SCI care.
  Interventions: Behavioral: Education (ED)

INTERVENTIONS:
Behavioral: Self Management (SM) — Self Management (SM) consists of: 1) on-site decisional support to promote provider adherence to ulcer management guidelines, 2) enhanced, interactive PrU education, 3) chronic disease self-management skill building via telephone based groups, 4) proactive care management using MI to support ongoing self-management activities, and 5) distance technology.
  Arms: SM+MI
Behavioral: Motivational Interviewing (MI) — Self Management and Motivational Interviewing (SM+MI) participants were assigned to both a self-management and motivational interview group. An education control intervention (ED) designed to be a credible intervention that is comparable to the SM will control for potential effects of natural history/time, treatment dosing, measurement processes, attention, the non-specific effects of therapeutic alliance, social support, and of receiving a manualized treatment with specific therapist procedures.
  Arms: SM+MI
Behavioral: Education (ED) — The ED intervention differs only in that subjects will not be instructed in any specific problem solving, self-monitoring, or SM techniques, with the exception of encouraging them to become informed consumers of SCI care.
  Arms: ED

SUMMARY:
Pressure ulcers (PrUs) are the most frequent significant medical complication after spinal cord injury (SCI). PrU prevalence, morbidity, mortality, and recurrence rates are high, and most persons with SCI will have at least one serious PrU during their lifetime. VA costs of treating the almost 3,500 unique Veterans with SCI and a severe ulcer at an SCI Center in FY10 was just under $400 million.

DETAILED DESCRIPTION:
Background:

Pressure ulcers (PrUs) are the most frequent significant medical complication after spinal cord injury (SCI). PrU prevalence, morbidity, mortality, and recurrence rates are high, and most persons with SCI will have at least one serious PrU during their lifetime. VA costs of treating the almost 3,500 unique Veterans with SCI and a severe ulcer at an SCI Center in 2010 was just under $400 million.

Objectives:

The primary objective of this randomized clinical trial (RCT) was to determine whether a multi-component self-management (SM) intervention increases the use of skin-protective behaviors and reduces skin worsening in Veterans with SCI, compared to an education control (ED) intervention. Secondary outcomes included PrU knowledge, self-management skills, communication with providers, self-efficacy, community integration and days on bedrest. Another objective was to conduct focus group interviews with patients and providers and to analyze transcripts of SM group sessions to determine barriers and facilitators with regard to spinal cord injury and pressure ulcer prevention.

Methods:

This was a multi-site efficacy intervention study with a single blind prospective randomized design. Descriptive statistics were used to summarize demographic and key variables. Supplemental focus group interviews were conducted with patients with SCI (n=35) and SCI providers (n=39). Focus group interviews and SM group calls were transcribed verbatim and analyzed using constant comparative techniques.

Study participants included Veterans hospitalized for Stage III/IV PrUs at or below the level of injury, from six VA SCI Centers around the country (Long Beach, Houston, Milwaukee, Augusta, Hines and St. Louis). Prior to discharge, PrU risk factors were identified and 1:1 PrU education was provided. Randomization and the behavioral interventions began at discharge. The number of randomized subjects were 72 in the ED group and 72 in the SM group (n=144). The analytic sample included subjects with complete data (n=92).

The intervention included 8 site coordinator-initiated calls using didactic (ED) or Motivational Interviewing (MI) strategies to address PrU risk factors. The second component included telephone group calls that included either didactic information about SCI or SM skills including: 1) knowledge about the medical condition; 2) self-monitoring; 3) problem-solving skills; 4) skill for managing the effects of the condition; 5) adherence to necessary health behaviors; and 6) self-advocacy with health care providers. ED subjects received general health information and were not instructed in any specific problem solving, self-monitoring or SM techniques. The ED intervention was comparable to the SM with respect to natural history/ time, dosing, measurement processes, attention, therapeutic alliance, social support, and in receiving a manualized treatment with specific therapist procedures. Self-reported outcome data were obtained by phone at 3 and 6 months, and from mailed photos of study ulcers.

Status:

Study is complete. Additional analyses are ongoing and future manuscripts are planned.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* SCI of at least six month's duration,
* hospitalized for a Stage III or IV PrU,
* cognitively intact,
* available for telephone follow-up, and
* discharged to a community setting or able to direct own care.

Exclusion Criteria:

We excluded patients with a terminal diagnosis, severe psychiatric comorbidities (eg, current psychosis), cognitive impairments that limited their ability to consent or participate, severe hearing loss, and wounds not expected to heal. People discharged to nursing homes unable to direct their own care were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marylou Guihan, PhD MA BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (5):
- United States (5):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

REFERENCES:
- [Result] Guihan M, Bombardier CH, Ehde DM, Rapacki LM, Rogers TJ, Bates-Jensen B, Thomas FP, Parachuri R, Holmes SA. Comparing multicomponent interventions to improve skin care behaviors and prevent recurrence in veterans hospitalized for severe pressure ulcers. Arch Phys Med Rehabil. 2014 Jul;95(7):1246-1253.e3. doi: 10.1016/j.apmr.2014.01.012. Epub 2014 Jan 30. PMID 24486242

RESULTS

PARTICIPANT FLOW:
Groups:
- Self Management (SM) + Motivational Interviewing (MI): Self Management (SM) + Motivational Interviewing (MI)
  Self Management and Motivational Interviewing (SM+MI): Self Management (SM) consists of: 1) on-site decisional support to promote provider adherence to ulcer management guidelines, 2) enhanced, interactive PrU education, 3) chronic disease self-management skill building via telephone based groups, 4) proactive care management using motivational interviewing to support ongoing self-management activities, and 5) distance technology.
- Education (ED): Education (ED)
  Education (ED): An education control intervention (ED) designed to be a credible intervention that is comparable to the SM will control for potential effects of natural history/time, treatment dosing, measurement processes, attention, the non-specific effects of therapeutic alliance, social support, and of receiving a manualized treatment with specific therapist procedures. The ED intervention will differ only in that subjects will not be instructed in any specific problem solving, self-monitoring, or SM techniques, with the exception of encouraging them to become informed consumers of SCI care.
Period: Overall Study
Arm/Group | Self Management (SM) + Motivational Interviewing (MI) | Education (ED)
Started | 72 | 72
Completed | 40 | 38
Not Completed | 32 | 34
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 22 | 26

BASELINE CHARACTERISTICS:
Population: For the SM+MI arm there was 1 death (post-randomization, pre-data collection) which accounts for the discrepency between starting participants (72) and baseline participants (71) for that group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Self Management (SM) + Motivational Interviewing (MI) | Education (ED) | Total
Number analyzed (Participants) | 71 | 72 | 143
Age, Continuous [Mean (Full Range); unit: years] | 59.4 [34 to 83] | 59.0 [22 to 85] | 59.3 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 69 | 70 | 139
Race/Ethnicity, Customized [Number; unit: participants]
  White | 46 | 52 | 98
  Black | 20 | 18 | 38
  Hispanic | 4 | 2 | 6
  Other | 1 | 0 | 1
Residence Type [Number; unit: participants]
  House | 50 | 56 | 106
  Apartment | 15 | 12 | 27
  Nursing Home | 1 | 0 | 1
  Other | 5 | 4 | 9
Marital Status [Number; unit: participants]
  Married | 29 | 28 | 57
  Never Married | 11 | 10 | 21
  Widowed | 5 | 6 | 11
  Divorced | 25 | 27 | 52
  Live with Partner | 0 | 1 | 1
  Missing | 1 | 0 | 1
Educational Level [Number; unit: participants]
  High School Graduate or Lower | 23 | 22 | 45
  Some College | 35 | 38 | 73
  College Graduate | 10 | 9 | 19
  Graduate School | 3 | 3 | 6
Duration of Spinal Cord Injury [Mean (Full Range); unit: years] | 23.8 [0.5 to 61.3] | 24.0 [0.5 to 60.9] | 24.0 [0.5 to 61.3]
Etiology [Number; unit: participants]
  Driving | 35 | 35 | 70
  Diving | 5 | 4 | 9
  Fall | 5 | 6 | 11
  Gunshot Wound | 6 | 11 | 17
  Other | 20 | 16 | 36
Level of Injury [Number; unit: participants]
  Cervical | 30 | 30 | 60
  Thoracic | 40 | 36 | 76
  Lumbar | 1 | 6 | 7
American Spinal Injury Association (ASIA) Score [Number; unit: participants] — The American Spinal Injury Association (ASIA) score is a scale to classify spinal cord injuries (SCI).
  A= complete SCI where no motor or sensory function is in the sacral segments S4-S5.
  B= incomplete SCI where sensory but not motor function is below the neurological level and includes the sacral segments S4-S5.
  C= incomplete SCI where motor function is below the neurological level and fewer than half of key muscles have a muscle grade < 3.
  D= incomplete spinal cord injury where motor function is below the neurological level and at least half of the key muscles have a muscle grade >3.
  participants
    A = Complete | 53 | 48 | 101
    B = Sensory Incomplete | 7 | 8 | 15
    C = Motor Incomplete | 7 | 10 | 17
    D = Motor Incomplete | 4 | 6 | 10
Source of Assistance [Number; unit: participants] — Participants can have more than one source of assistance.
  participants
    Spouse; partner/significant other; Relative | 50 | 45 | 95
    Paid Attendant | 30 | 18 | 48
    Other Regular Assistance | 5 | 8 | 13
    No Regular Assistance | 12 | 11 | 23
Comorbid Conditions (baseline) [Number; unit: participants]
  Diabetes | 34 | 22 | 56
  Depression | 29 | 29 | 58
  Osteomyelitis | 18 | 10 | 28
Salzburg PrU Risk Score [Mean (Full Range); unit: Scores on a scale] — The Salzberg PrU risk scale was developed as a pressure ulcer risk assessment scale specifically for persons with SCI using a list of identified risk factors contributing to PrU development. Total individual scores range from 0 to 25, with a higher score indicating a greater risk of developing a PrU.
  Salzberg, C. Andrew, et al. "A New Pressure Ulcer Risk Assessment Scale for Individuals With Spinal Cord Injury." American Journal of Physical Medicine & Rehabilitation 75.2 (1996): 96-104.
  Scores on a scale | 9.8 [4 to 18] | 9.3 [5 to 17] | 9.5 [4 to 18]
Pressure Ulcer (PrU) Characteristics [Mean (Full Range); unit: Pressure Ulcers]
  Number of prior PrUs | 2.89 [0 to 25] | 1.93 [0 to 8] | 2.41 [0 to 25]
  Number of current PrUs | 1.6 [1 to 5] | 1.3 [1 to 3] | 1.4 [1 to 5]
PrU Size of Largest Ulcer [Mean (Full Range); unit: cm^2] | 8.2 [0.1 to 39.1] | 4.5 [0.1 to 22.0] | 6.3 [0.1 to 39.1]
PrU Duration for Largest PrU [Mean (Standard Deviation); unit: days] | 213 (244) | 407 (631) | 307 (482)
Prior PrU Surgery [Number; unit: participants]
  Yes | 51 | 46 | 97
  No | 20 | 26 | 46
History of PrUs [Number; unit: participants] | 56 | 56 | 112
Locations of Current Pressure Ulcers [Number; unit: Pressure Ulcers] — Patients can have more than one ulcer present at randomization
  Pressure Ulcers
    Ischium | 40 | 38 | 78
    Trochanter | 11 | 9 | 20
    Sacrum | 15 | 13 | 28
    Coccyx | 9 | 6 | 15
    Other locations (e.g., feet) | 16 | 16 | 32
Stage of PrUs at randomization [Number; unit: Pressure Ulcers] — Patients can have more than one ulcer present at randomization. Stage III: Full thickness tissue loss. Subcutaneous fat may be visible but bone, tendon, or muscle are not exposed. Slough may be present but does not obscure the depth of tissue loss. May include undermining and tunneling.
  Stage IV: Full thickness tissue loss with exposed bone, tendon, or muscle. Slough or eschar may be present on some parts of the wound bed. Often includes undermining and tunneling.
  Pressure Ulcers
    Stage III = Full thickness | 22 | 31 | 53
    Stage IV = Full thickness | 54 | 43 | 97
Hospital-acquired PrU [Number; unit: Pressure Ulcers] | 12 | 9 | 21
Current Employment [Number; unit: participants]
  Unemployed | 60 | 61 | 121
  Employed | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percent of Possible Self-Reported Skin Care Behaviors
Description: Skin Behavior Change was calculated as the percentage of Self-Reported Behavior at 3 and 6 months (minus the percentage at baseline).
  The study reported the number of guideline-recommended skin care behaviors, assessed by the Skin Care Behavior Checklist, a self-reported measure of adherence to 8 guideline recommended skin care behaviors. The average percentage of the 8 behaviors adhered to for each participant was measured by intervention arms at admission (baseline), 3 and 6 months post-discharge.
Time Frame: Admission (Baseline), 3 months, 6 months
Measure: Mean (Standard Deviation); unit: % of Possible Self-Reported Behaviors
Arm/Group | Self Management (SM) + Motivational Interviewing (MI) | Education (ED)
Number analyzed (Participants) | 71 | 72
% of Possible Self-Reported Behaviors
  Admission | 73.8 (23.3) | 74.1 (18.6)
  3 Months | 83.5 (17.5) | 79.5 (19.6)
  6 Months | 85.0 (15.2) | 83.0 (14.6)

2. Primary Outcome: Skin Behavior Change
Description: Self-reported improvement in skin care behaviors in the SM+MI versus ED control intervention arms.
  The study reported the number of guideline-recommended skin care behaviors, assessed by the Skin Care Behavior Checklist, a self-report measure of adherence to 8 skin care behaviors for each participant.The difference in the average percentage of the 8 behaviors adhered to by each participant was measured for the different intervention arms from admission (baseline) to 3 and 6 months post-discharge.
Time Frame: Admission (Baseline), 3 months, 6 months
Measure: Mean (Standard Deviation); unit: % Change
Arm/Group | Self Management (SM) + Motivational Interviewing (MI) | Education (ED)
Number analyzed (Participants) | 71 | 72
% Change
  Baseline to 3 months | 9.7 (19.3) | 5.4 (22.9)
  Baseline to 6 months | 11.3 (20.0) | 8.9 (18.1)

3. Primary Outcome: Any Skin Worsening
Description: Skin worsening was defined as when a participant with an open wound at the time of discharge is found to have >20% wound area at 3 or 6 months post-discharge (including new wounds and reopened wounds). Worsening was also defined as a when a participant with a closed wound at discharge is found to have a new or reopened wound at 3 or 6 months post-discharge.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Self Management (SM) + Motivational Interviewing (MI) | Education (ED)
Number analyzed (Participants) | 71 | 72
participants
  No | 36 | 33
  Yes | 35 | 39

4. Primary Outcome: Skin Status
Description: as for outcome 3
Time Frame: Admission (Baseline), 3 months, 6 months
Measure: Number; unit: participants
Arm/Group | Self Management (SM) + Motivational Interviewing (MI) | Education (ED)
Number analyzed (Participants) | 71 | 72
participants
  No Skin Worsening | 36 | 33
  Worse 0-3 Months | 26 | 28
  Worse 4-6 Months | 9 | 11

5. Secondary Outcome: Mean Number of Skin-related Admissions
Description: Post-discharge skin-related hospitalizations were for both groups (SM+MI vs. ED) but not as study-related or as an adverse event. This study examined an outpatient intervention during which rehospitalization could be triggered by the participants' early reporting of skin breakdown.
Time Frame: Discharge to end of study (6 months)
Population: Mean number of skin-related post-discharge admissions (ICD9 code =707.xx)
Measure: Mean (Standard Deviation); unit: admissions/participant
Groups:
- SM+MI Group: Self Management (SM) + Motivational Interviewing (MI). Motivational Interviewing (MI) is an evidence-based form of counseling to improve behavior change. Self Management (SM) includes: 1) ulcer management guidelines, 2) enhanced, interactive PrU education, 3) chronic disease self-management skill building via telephone based groups, 4) proactive care management using MI to support ongoing self-management activities, and 5) distance technology.
- ED Group: An education control intervention (ED) designed to be a credible intervention that is comparable to the SM will control for potential effects of natural history/time, treatment dosing, measurement processes, attention, the non-specific effects of therapeutic alliance, social support, and of receiving a manualized treatment with specific therapist procedures. The ED intervention will differ only in that subjects will not be instructed in any specific problem solving, self-monitoring, or SM techniques, with the exception of encouraging them to become informed consumers of SCI care.
  The ED intervention differs only in that subjects will not be instructed in any specific problem solving, self-monitoring, or SM techniques, with the exception of encouraging them to become informed consumers of SCI care.
Arm/Group | SM+MI Group | ED Group
Number analyzed (Participants) | 72 | 72
admissions/participant | 1.5 (0.8) | 1.6 (0.7)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Self Management (SM) + Motivational Interviewing (MI) | Education (ED)
Serious Adverse Events (participants affected / at risk) | 4/72 | 3/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self Management (SM) + Motivational Interviewing (MI) (N=72) | Education (ED) (N=72)
Death (Investigations) | 4 (4) | 3 (3) — Cause of death was not systematically tracked throughout study, and deaths were unrelated to the study intervention.

LIMITATIONS AND CAVEATS:
The study was underpowered because of difficulties encountered with recruitment and retention. Delivering an adequate "dose" of the treatments and site coordinator fidelity to the MI intervention were also limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes